CLINICAL TRIAL: NCT05968300
Title: Getting INFORMED and Living Well: A Demonstration Project to Facilitate Pandemic Recovery Among Asian Americans in California
Brief Title: Getting INFORMED and Living Well Among Asian Americans in California
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Chinese Community Health Resource Center (Other); University of California, Davis (Other); University of California, Merced (Other); California Department of Public Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P0567396
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; Well-Being, Psychological
Keywords: Asian Americans; Peer Education; Immigrants; Chinese; Hmong; Korean; Vietnamese
MeSH Terms: conditions — COVID-19; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Non-randomized trial (Preference trial)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INFORMED-Living Well (Experimental): INFORMED-Living Well consists of two components: 1) LHW outreach support providing responsive education and support; and 2) a 6-week automated SMS text messaging. The LHW educational outreach component includes 2 small group educational sessions with 2-8 participants. Participants will also receive a weekly SMS Text or instant message on managing emotional wellness within and beyond the context of the COVID-19 pandemic over 6 weeks. In addition, participants will receive as-needed messages on updates of COVID-19 or other situations that may introduce new worries and tragic culturally-based traumatic events.
  Interventions: Behavioral: INFORMED-Living Well
- Text Messaging Only (Active Comparator): Participants will have a 6-week SMS text messaging program identical to that received by the INFORMED-Living Well participants.
  Interventions: Behavioral: Text Messaging Only

INTERVENTIONS:
Behavioral: INFORMED-Living Well — 1) LHW outreach support providing responsive education and support; and 2) a 6-week automated SMS text messaging
  Arms: INFORMED-Living Well
Behavioral: Text Messaging Only — A 6-week automated SMS text messaging
  Arms: Text Messaging Only

SUMMARY:
The project is to facilitate pandemic recovery by promoting emotional wellness among Asian Californians. The intervention includes a 6-week program in which participants may choose to receive text only or text + Lay Health Worker outreach targeting 600 self-identified Asian Americans residing in California who speak/read English, Chinese, Korean, Hmong, or Vietnamese.

DETAILED DESCRIPTION:
Investigators will conduct a non-randomized intervention trial (preference trial). Research participants involved in the trial will include 20 lay health workers (LHWs) and 600 trial participants with intervention delivered via SMS text messaging (for all participants), and the intervention group will receive educational intervention outreach from an LHW via Zoom or mutually agreed video conferencing online venues, and by telephone or instant messaging. Participants will choose which group they are in, SMS text messaging only or SMS text messaging plus educational outreach from an LHW.

ELIGIBILITY:
Inclusion Criteria:

i) age 18 and older

ii) speak Chinese, English, Hmong, Korean, or Vietnamese

iii) self-identify as Asian American

iv) have access to a mobile phone to receive SMS text messages

Exclusion Criteria:

* unwilling to receive SMS text messages from the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change in decisional conflict scale (SURE) scores | Baseline and 8-week follow-up
  Self-assessed perceptions of decision conflict will be assessed using the 4-item Decision Conflict Scale (SURE). Scores on the SURE scale range from 0 to 4, with higher scores indicating less decisional conflict. A score of less than 4 indicates decisional conflict.

SECONDARY OUTCOMES:
Change in proportion of participants who have Intention to seek help for mental health | Baseline and 8-week follow-up
  We will use a survey item to assess participants' intention to seek help for mental health issues when needed. A response will be 0 (No) or 1 (Yes).
Change in self-reported emotional wellness outcome | Baseline and 8-week follow-up
  We will use the four-item Patient Health Questionnaire (PHQ4) for measuring anxiety and depression symptoms. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12). Total score 3 or higher for the first 2 questions suggests anxiety, and total score 3 or higher for the last 2 questions suggests depression.
Change in the percentage of participants' awareness of resources to get help or to learn more about improving emotional wellness | Baseline and 8-week follow-up
  We will assess participants' awareness of resources to get help or to learn more about improving emotional wellness. Two items created for the study will be used: 1) Do you know about "988"? (Yes, No, Unsure) 2) Do you know where to get help for mental health issues when you need to? (Yes, No, Unsure). The percentage of participants who answer "yes" to both questions will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - The Fresno Center, Fresno, California
  - Chinese Community Health Resource Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Immigrant Resettlement & Cultural Center, San Jose, California

IPD SHARING:
Plan to Share IPD: No